CLINICAL TRIAL: NCT04879082
Title: Identification of Occupational Exposures in Patients With Interstitial Lung Diseases (ILD)
Brief Title: Identification Of Occupational Exposures In Patients With ILD
Acronym: ILD
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: A257
Record Dates: First submitted 2021-03-26; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-03

CONDITIONS: Occupational Exposure; Interstitial Lung Disease
Keywords: Occupational Exposure; Lung Fibrosis; Interstitial Lung Disease; Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — Occupational Exposure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ILD: Patients with ILD, whose file has been discussed in a multidisciplinary meeting since May 2020 at the Louis Pradel Pneumological Hospital, and who have benefited from a professional interview in the Occupational pathology consultation center of the Hospital Center Lyon Sud.
  Interventions: Other: Professional course, occupational exposures

INTERVENTIONS:
Other: Professional course, occupational exposures — The data collected are the following variables: age, sex, diploma, professional course coded in CITP (International Standard Classification of Professions) and NAF (French Nomenclature of Activities), occupational exposures, smoking, risk factors non-professionals, clinical elements of ILD and elements relating to an occupational disease certificate. This database is anonymized.
  The precise diagnosis of ILD is retained during the multidisiciplinary meeting.
  Occupational exposures are assessed in specialized consultation :
  * a first professional interview phase: The professional history is traced, listing the training courses followed and the trades carried out. The questioning is precise and focuses on the different tasks performed, and the products used.
  * a second step, where a questionnaire is completed by the doctor: A list of specific substances is offered to the patient, who responds whether or not he thinks he has been exposed to them in his professional past.

SUMMARY:
Diffuse interstitial lung disease brings together a heterogeneous group of pulmonary pathologies, characterized by infiltrating and diffuse lesions of the pulmonary interstitium. The evolving risk of these ILD is pulmonary fibrosis, with the development of chronic respiratory failure.

The process of the etiological diagnosis of ILD results from a multidisciplinary approach (pulmonologists, radiologists, occupational health specialists, anatomo-pathologists, etc…). Indeed, the multitude of possible causes of these diseases makes the etiological diagnosis difficult. Professional aetiologies are also frequently mentioned : pneumoconiosis, hypersensitivity pneumonitis, as a differential diagnosis.

It therefore appears essential to deepen the professional aspect during the diagnostic process for ILD.

Since May 2020, a professional interview has been systematically offered by the Occupational Pathology Consultation Center of the Hospital Center Lyon Sud, to patients followed by the team of Professor Vincent COTTIN, whose file was discussed in a multidisciplinary meeting.

The data collected to constitute a database are the following variables: age, sex, diploma, professional course coded in CITP (International Standard Classification of Professions) and NAF (French Nomenclature of Activities), occupational exposures, smoking, risk factors non-professionals, clinical elements of ILD and elements relating to an occupational disease certificate. This database is anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ILD.
* File discussed in a multidisciplinary meeting since May 2020 at the Louis Pradel Pneumological Hospital.
* Have benefited from a professional interview in the Occupational pathology consultation center of the Hospital Center Lyon Sud.

Exclusion Criteria:

* Patients with sarcoidosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ILD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Study the distribution of occupational exposures according to the types of ILD. The precise diagnosis is retained during the multidisiciplinary meeting. | The precise diagnosis of ILD is retained immediately after the multidisiciplinary meeting.
  Precise diagnosis of ILD : type of PID diagnosed
Occupational exposures are assessed in specialized consultation by the occupational physician. | Occupational exposures are assessed immediately after the occupational consultation.
  Occupational exposures

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de consultation de pathologie professionnelle, Centre Hospitalier Lyon Sud, Pierre-Bénite, France